CLINICAL TRIAL: NCT07344688
Title: Effect of White Tea (Camellia Sinensis L.) Beverages on Anthropometric, Hematological, Biochemical and First Line Antioxidant Enzymes Activity of Healthy Human (Superoxide Dismutase, and Glutathione Peroxidase)
Brief Title: The Effect of White Tea in Healthy Human Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PHAR.202509-01
Record Dates: First submitted 2025-09-12; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Healhty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- White tea intervention (Experimental): Nineteen respondents will be given 200 mL of white tea (4 grams of white tea sample in 200 mL of water at a temperature of 95-98°C) for 14 days after a 7-day washout period. In the final stage, all respondents will undergo an observation phase. In the final stage, all respondents are required to submit updates on their physical condition. If they experience discomfort such as nausea, dizziness, or general unease, the respondents will be examined by the research physician. In our study, no control group was used. To demonstrate the effect of white tea on the respondents' health condition, we compared the results before and after the treatment.
  Interventions: Other: White tea intervention

INTERVENTIONS:
Other: White tea intervention — 1. White tea infusion was prepared by brewing 4 grams of white tea in 200 mL of hot water.
  2. Healthy respondents were asked to consume the white tea infusion for 14 days.
  3. The focus of this study was to observe the effect of white tea infusion on antioxidant enzyme activity and its relationship with anthropometric, biochemical, and haematological parameters.

SUMMARY:
This clinical study aims to determine the effects of consuming white tea infusion (Camellia sinensis) on healthy subjects over a period of 14 days. The main questions it aims to answer are:

1. Determine the effect of white tea consumption on the anthropometry of healthy subjects.
2. Determine the effect of white tea consumption on the biochemical parameters of healthy subjects.
3. Determine the effect of white tea consumption on hematology parameters that are related to anemia case in healthy subjects.
4. Determine the effect of white tea consumption on the activity of first-line antioxidant enzymes in healthy subjects

Researchers used only one treatment group, and respondents knew which treatment they would receive (single-arm and open-labelled), namely white tea infusion to maintain human body health. Participants will:

1. Follow the washout stage for 7 days
2. Drink white tea infusion every day for 14 days.
3. Follow up to monitor adverse effects after consuming white tea; this stage will be conducted for 7 days.
4. Report all food and beverages consumed by respondents during the study.

DETAILED DESCRIPTION:
Unhealthy lifestyles, including alcohol consumption, illegal drug use, radiation exposure, and the preparation of food (e.g. smoked meat, used oil, and fat) and polluted environments (water and air pollution) are triggering an increase in cases of degenerative diseases worldwide, including ischaemic heart disease, diabetes, cancer, atherosclerosis, liver disease, kidney disease, chronic obstructive pulmonary disease, and others. The body's natural defences can decline at any time due to the development of reactive oxygen species (ROS) caused by unhealthy lifestyle factors and environmental pollution. Exogenous antioxidants are important for maintaining the body's defence system against excessive ROS. This study will examine the potential of compounds in white tea infusion in maintaining human health by monitoring several parameters, including anthropometric, biochemical, haematological, and antioxidant enzyme activity. The anthropometric parameters tested include body weight, height, waist circumference, systolic blood pressure, and diastolic blood pressure. Biochemical parameters include lipid profile (total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides), alanine aminotransferase (ALT), aspartate aminotransferase (AST), serum creatinine levels, estimated glomerular filtration rate (eGFR), and urea nitrogen levels. The haematological parameters used are directly related to the indication of anaemia, including red blood cell count, haemoglobin, haematocrit, mean corpuscular haemoglobin (MCH), and mean corpuscular volume (MCV). Finally, there are the first-line antioxidant enzyme activity parameters, including superoxide dismutase (SOD), catalase (CAT), and glutathione peroxidase (GPx). This examination was conducted before and after the 14-day white tea infusion treatment to observe the effects of the treatment. Male and female healthy volunteers were instructed to follow three stages of research, including:

1. Washout phase : respondents are advised to avoid products with high polyphenol content such as turmeric, ginger, galangal, grapes, apples, oranges, coffee, other types of tea, and chocolate, either directly or in processed products.
2. Treatment phase: respondents continue to avoid the products avoided during the washout process. In this phase, respondents will consume white tea infusion (4 grams of WT in 200 mL of freshly boiled water) every day for 14 days.
3. Observational phase: the phase is conducted for 7 days to monitor the presence or absence of side effects after 14 days of consuming white tea infusion.

ELIGIBILITY:
Inclusion Criteria:

1. The participants are the community around Padjadjaran University with an age range of 20 - 35 years old. Female respondents were unmarried.
2. The participants are non-smoker.
3. The participants should have no history of anemia, chronic disease, hepatic and renal dysfunction.
4. The participants are willing to follow the research process until its finish by signing an informed consent form.

Exclusion Criteria:

1. The participants who are undergoing drug therapy and taking vitamin supplements.
2. The participants who failed due to illness or are unable to continue the examination to the end.
3. Respondents with pre-treatment biochemical results not within the normal range

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Antioxidant Enzymes Analysis | 14 days
  Comparing the antioxidant activity values of enzymes including superoxide dismutase, catalase, and glutathione peroxidase in pre and post white tea treatment (day 0 and day 15). The increased activity of antioxidant enzymes signifies an enhancement in the body's capability to combat free radicals. The analysis will be conducted using a reagent kit to obtain the antioxidant enzyme activity values in the respondents' serum. All antioxidant enzyme parameter values are expressed in U/mL.
Liver Function Analysis | 14 days
  The effect of the product on liver function will be analysed based on SGOT and SGPT values. A drastic increase compared to the pre-intervention level indicates potential toxicity. Both parameters will be expressed in units of ukat/L.
estimated Glomerular filtration rate | 14 days
  A drastic decrease in eGFR indicates the potential toxicity of white tea beverages. eGFR results of respondents will be expressed in mL/min/1.73m2
Lipid profile measurement | 14 days
  The effect of product administration on lipid profile was assessed by measuring total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL) parameters. Product effectiveness was determined based on the stability or decrease in total cholesterol, triglycerides, and LDL values, as well as an increase in HDL values post-treatment compared to pre-treatment values. Total cholesterol, triglycerides, low-density lipoprotein (LDL), and high-density lipoprotein (HDL) will be expressed in mmol/L
Fasting blood glucose measurement | 14 days
  Fasting blood glucose will be expressed in mmol/L
Serum creatinine Analysis | 14 days
  An elevated serum creatinine level is an indication of potential toxicity associated with white tea consumption. Serum creatinine level will be expressed in umol/L
Blood Urea Nitrogen Analysis | 14 days
  An elevated blood urea nitrogen level is an indication of potential toxicity associated with white tea consumption. The parameter will be written in units of mmol/L

SECONDARY OUTCOMES:
Body Weight Measurement | 14 days
  The body weight of respondents will be measured on day 0 and day 15 after administration of white tea treatment. Body weight values before and after treatment will be analysed. Body weight values will be recorded in kilograms (kg)
Body Height Measurement | 14 days
  Height measurements will be taken on days 0 and 15. Measurements will be taken to calculate BMI values for further analysis. Height values will be recorded in centimetres (cm).
Body Mass Index | 14 days
  Body mass index measurements will be taken using weight and height data. The BMI result is recorded in kg/m^2, then the analysis will be classified into the categories of underweight (BMI range <18.5 kg/m^2) healthy (BMI range 18.5 - 24.9 kg/m^2), overweight (BMI range 25.0 - 29.9 kg/m^2) and obese (BMI range > 29.9 kg/m^2).
Waist Circumference Measurement | 14 days
  Waist circumference measurements were taken on days 0 and 15 using a measuring tape and expressed in centimetres (cm). The results before and after treatment will be analysed.
Blood Pressure Measurement | 14 days
  Both systolic blood pressure or diastolic blood pressure will be measured.
Number of participants with serious adverse events related to study product | 14 days
  Signs and symptoms of adverse event related to study product including nausea, vomiting, dizziness, burning sensation in the stomach, excessive fatigue, constipation, and excessive urination will be assessed daily for 14 days since the first administration of white tea beverages.
Red Blood Cells Measurement | 14 days
  Red blood cell (RBC) parameters are one of the parameters used to assess whether white tea beverages have the potential to cause anaemia. Tests were conducted on days 0 and 15, the difference in RBC values was analysed, and RBC values were expressed in 10^6/uL.
Haemoglobin Measurement | 14 days
  Haemoglobin parameters are one of the parameters used to assess whether white tea beverages have the potential to cause anaemia. Tests were conducted on days 0 and 15, the difference in haemoglobin values was analysed, and haemoglobin values were expressed in grams/decilitre (g/dL)
Haematocrit Measurement | 14 days
  Haematocrit parameters are one of the parameters used to assess whether white tea beverages have the potential to cause anaemia. Tests were conducted on days 0 and 15, the difference in haematocrit values was analysed, and haematocrit values were expressed in percentage (%).
Mean Corpuscular Haemoglobin Measurement | 14 days
  Mean Corpuscular haemoglobin (MCH) parameters are one of the parameters used to assess whether white tea beverages have the potential to cause anaemia. Tests were conducted on days 0 and 15, the difference in MCH values was analysed, and MCH values were expressed in picograms (pg).
Mean Corpuscular Volume Measurement | 14 days
  Mean Corpuscular Volume (MCV) parameters are one of the parameters used to assess whether white tea beverages have the potential to cause anaemia. Tests were conducted on days 0 and 15, the difference in MCV values was analysed, and MCV values were expressed in femtoliters (fL).
Daily intake | 28 days
  The daily report of respondents incorporates information regarding their daily activities and the consumption of food and beverages during the 28-day research period. Respondents will be asked to submit this data every day via personal chat (WhatsApp).

CONTACTS AND LOCATIONS:
Overall Officials: Gofarana Wilar, Ph.D., Study Director — Faculty of Pharmacy, Universitas Padjadjaran, Bandung, Indonesia
Locations (1):
- Faculty of Pharmacy, Padjadjaran University, Sumedang, West Java, Indonesia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2026-01-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT07344688/Prot_SAP_000.pdf